CLINICAL TRIAL: NCT03677258
Title: Non-interventional Study: Collagen Anti-age Treatment in Routine Clinical Practice
Brief Title: Effectiveness and Safety of Collagen Complex COLLOST in Anti-age Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nearmedic Plus LLC (Industry)
Collaborators: Institute of Plastic Surgery and Cosmetology, Moscow, Russia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLLOST postmarketing study
Record Dates: First submitted 2018-04-25; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Skin Aging
Keywords: Collagen; anti-age therapy; cosmetology; lifting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen injections (Experimental): 30 females with aging facial problems from 35 to 65 years old prescribed collagen ingection once every 3 weeks, cours of therapy - 3 procedures
  Interventions: Device: Collagen for injections 7%
- Hyaluronic acid injections (Active Comparator): 30 females with aging facial problems from 35 to 65 years old prescribed hyaluronic acid ingection once every 3 weeks, cours of therapy - 3 procedures
  Interventions: Device: Hyaluronic acid for injections 2%

INTERVENTIONS:
Device: Collagen for injections 7% — Injection of medical device
  Other Names: Collost
  Arms: Collagen injections
Device: Hyaluronic acid for injections 2% — Injection of medical device
  Other Names: Viscoderm
  Arms: Hyaluronic acid injections

SUMMARY:
This study evaluates the statistics of anti-age treatment in outpatient sites in Russia (involution indicators: clinical scales; instrumental diagnostics, ultrasonic scannings, assesment of allergic state, efficacy assesment in according with GAIS scale) in routine clinical practice with focus on collagen therapy.

DETAILED DESCRIPTION:
This non-interventional study covers 60 patients (females with involuntary changes of the face skin) from Russian sites.

The following data will be collected and analyzed after the end of treatment:

* demography
* assessment of allergic state
* safety data
* severity of aging effect
* clinical scales results before 1visit and after end of treatment
* GAIS effectiveness assessment
* instrumental diagnostic before 1visit and after end of treatment
* hydration
* elasticity
* microcirculation level
* lipofuscin level
* ultrasound scanning
* derma echo density

ELIGIBILITY:
Inclusion Criteria:

* signed Inform Consent Form
* only females
* from 35 to 65 years old
* 1-3 skin photo types
* signs of age-related skin changes
* absence of chronic disease in decompensation phase
* refusal to receive any cosmetic procedures during the study

Exclusion Criteria:

* pregnancy, lactation period
* infection process, dermatoses, censers
* systemic connective tissue diseases with skin and subcutaneous tissue damage
* taking isotretinoin drugs for the previous 6 months
* propensity to form hypertrophic and keloid scars
* exacerbation or decompensation of chronic somatic diseases; infectious and oncological diseases
* violations of blood coagulation, including iatrogenic (taking drugs that affect blood clotting)
* taking antihistamines, glucocorticoids, NSAIDs, immunosuppressants and other drugs that affect the reactivity of the skin
* hypersensitivity to the components of the studied medical device

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Anti-aging therapy more popular for female patients
Enrollment: 60 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
Elastisity Ultrasonic scanning of the scin - epidermis and dermis in 3 area of the face after injections of the Collagen and after injections of the Hyaluronic Acid | 3 months
  To evaluate elasticity in Cheek, in forehead and glabella area scanned after each procedure and compare with screening results

SECONDARY OUTCOMES:
Safety: to evaluate safety by comparing adverse events after injections of the Collagen and after injections of the Hyaluronic Acid | 3 months
  To evaluate safety by comparing adverse events and their relationships with medical devices
Microcirculation data after injections of the Collagen and after injections of the Hyaluronic Acid | 3 months
  To evaluate results after each procedure and after 3 procedures by the laser Doppler fluorimetry
3D photo materials after injections of the Collagen and after injections of the Hyaluronic Acid | 3 months
  To evaluete results of procedures by the Quantifirecare data
GAIS scale data after injections of the Collagen and after injections of the Hyaluronic Acid | 3 months
  To evaluete results of 1 procedures and after 3 procedures by the patient and by the doctor

CONTACTS AND LOCATIONS:
Overall Officials: Anna Stenko, PhD, Principal Investigator — Institute of Plastic Surgery and Cosmetology
Locations (1):
- Institute of Plastic Surgery and Cosmetology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided